CLINICAL TRIAL: NCT07203248
Title: A Real-world Study on the Use of CGRP-targeted Medications for the Treatment of Vestibular Migraine in Chinese Patients
Brief Title: Chinese Real-world Study of Treatment of Vestibular Migraine
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First People's Hospital of Hangzhou (Other); Sir Run Run Shaw Hospital (Other); Affiliated Hospital of Jiaxing University (Other); The People's Hospital of Quzhou (Other); The First People Hospital of Hangzhou Lin An District (Unknown); Shaoxing People's Hospital (Other); Jiaxing Hospital of T.C.M (Unknown); Hangzhou Hospital of Traditional Chinese Medicine (Other); Affiliated Wenling Hospital of Wenzhou Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); The First People's Hospital of Huzhou (Other); Xin Hua Hospital of Zhejiang Province (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Huzhou Central Hospital (Other); Chinese Medical University (Unknown); Tiantai People Hospital (Unknown); Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 20250455
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Vestibular Migraine; Dizziness; Vertigo
Keywords: Vestibular Migraine; CGRP; acute treatment; preventive treatment; real-world
MeSH Terms: conditions — Dizziness; Vertigo | interventions — Calcitonin Gene-Related Peptide Receptor Antagonists

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- A1: Group A is the acute treatment group, which will observe the effectiveness of medication used for acute treatment after a VM (Vestibular Migraine) attack in the participants. Subgroup A1 will include participants who undergo acute treatment with CGRP-targeted drugs.
  Interventions: Drug: CGRP R Inhibitor; CGRP Inhibitor
- A2: Group A is the acute treatment group, which will observe the effectiveness of medication used for acute treatment after a VM (Vestibular Migraine) attack in the participants. Subgroup A2 will include participants who undergo acute treatment with medications other than CGRP drugs (such as NSAIDs, triptans, etc.).
  Interventions: Drug: none-CGRP
- B1: Group B is the preventive treatment group, which will observe the efficacy of 12-week prophylactic medication in participants. Subgroup B1: Patients receiving CGRP-targeted drugs (e.g., CGRP monoclonal antibodies or gepants) for preventive treatment.
  Interventions: Drug: CGRP R Inhibitor; CGRP Inhibitor
- B2: Group B is the preventive treatment group, which will observe the efficacy of 12-week prophylactic medication in participants. Subgroup B2: Patients receiving non-CGRP preventive medications (e.g., flunarizine, topiramate, propranolol, etc.).
  Interventions: Drug: none-CGRP

INTERVENTIONS:
Drug: CGRP R Inhibitor; CGRP Inhibitor — Participants who are prescribed CGRP class drugs for the acute treatment of VM will be considered for inclusion in Group A1.Participants who are prescribed CGRP class drugs for the preventive treatment of VM will be considered for inclusion in Group B1.
  Groups: A1; B1
Drug: none-CGRP — Participants who are prescribed none-CGRP class drugs for the acute treatment of VM will be considered for inclusion in Group A2.Participants who are prescribed none-CGRP class drugs for the preventive treatment of VM will be considered for inclusion in Group B2.
  Groups: A2; B2

SUMMARY:
Vestibular migraine is a phenotype of migraine, characterized by more prominent vertigo symptoms compared to headache. Treatments for VM are mainly divided into two categories: acute treatment and preventive treatment. Acute treatment aims to reduce the severity and duration of a single episode, while preventive treatment aims to decrease the frequency, severity, and duration of attacks. Current acute treatments are primarily divided into pain relief and anti-dizziness, with specific drugs such as triptans and ergots being applicable for pain relief, but only betahistine has weak evidence for anti-dizziness, and relevant clinical evidence is very scarce. Preventive treatment mainly refers to migraine preventive treatments, with recommended medications including traditional drugs like topiramate, flunarizine, propranolol, etc., but the efficacy and safety of these drugs are limited. CGRP-targeted drugs are believed to play a role in the preventive treatment of VM, and there are related literature reports, but most are small-sample studies or retrospective studies. This study aims to explore the real-world efficacy of CGRP-targeted drugs in the acute and preventive treatment of VM through a prospective real-world study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 75 years.
2. Meet the following criteria established by the Barany Society for the diagnosis of vestibular migraine or probable vestibular migraine:

   Vestibular Migraine A: At least five episodes with moderate or severe vestibular symptoms lasting from 5 minutes to 72 hours.

   B: Current or past history of migraine, with or without aura, according to the International Classification of Headache Disorders (ICHD-3).

   C: One or more migraine features during at least 50% of vestibular episodes:

   Headache with at least two of the following characteristics: unilateral, pulsating, moderate or severe pain, worsening with routine physical activity.

   Photophobia and phonophobia. Visual aura. D: Not better accounted for by another vestibular or ICHD diagnosis. Probable Vestibular Migraine A. At least five episodes with moderate or severe vestibular symptoms lasting from 5 minutes to 72 hours.

   B. Meets only one of the criteria B or C for vestibular migraine (history of migraine or migraine features during episodes).

   C. Not better accounted for by another vestibular or ICHD diagnosis.
3. More than or equal to 4 days per month with confirmed vestibular symptom in the three months prior to enrollment (only required for group B).
4. Able to complete at least 80% of the electronic diary during the treatment period.
5. The investigator believes that the participant is able to read, understand, and complete the study questionnaires and headache diary.

Understanding and compliance with the study procedures and methods, voluntary participation in this trial, and written informed consent.

Exclusion Criteria:

1. Pregnant women, breastfeeding women, or those unwilling to use approved contraceptive methods during study participation.
2. Presence of a condition or abnormality that the investigator believes would affect the safety of the patient or the quality of the data.
3. History of ear surgery (excluding ear tube surgery).
4. Other vestibular diagnoses (excluding treated benign paroxysmal positional vertigo, BPPV). This includes Ménière's disease, superior semicircular canal dehiscence syndrome, vestibular neuritis, persistent postural-perceptual dizziness, unilateral or bilateral vestibular hypofunction, cerebellar or brainstem disorders, multiple sclerosis, or seasickness.
5. More than two preventive migraine medications have failed.
6. Previous or current treatment with CGRP class drugs.
7. History of serious medical or psychiatric conditions, as judged by the treating physician (including significant coronary artery disease, peripheral vascular disease, cerebrovascular disease, renal disease, liver disease, Raynaud's disease, uncontrolled psychiatric illness, or past psychiatric hospitalization).
8. History of mania, psychosis, or suicidal ideation.
9. Acceptable if using no more than two migraine preventive medications (prescribed specifically for this purpose), with stable dosing for at least 2 months prior to study start.
10. History of drug or alcohol abuse within the 12 months prior to screening, based on the participant's medical records or self-report.
11. Those who have received or plan to receive botulinum toxin (e.g., Dysport®, Botox®, Xeomin®, Myobloc®, Jeuveau™) for therapeutic or cosmetic purposes in the head, face, or neck within 4 months prior to screening or during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will recruit male and female participants aged 18 to 75 years in China, who have vestibular migraine diagnosed according to the VM definition published by the Bárány Society in 2012. Participants must be prescribed with CGRP class drugs based on the clinical judgment of the physician and the willingness of the participants. Participants in Groups A1 and B1 will be considered for screening for eligibility criteria only after being prescribed with CGRP class drugs. Participants in Groups A2 and B2 will be considered for screening for eligibility criteria only after being prescribed with non-CGRP class drugs.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The average scores of the most severe vestibular symptom post-dose measured by VAS scale to evaluate the effectiveness of CGRP medication in the acute treatment of vestibular migraine | within 48 hours post-dose of CGRP medication
  Vestibular symptom severity post-dose will be measured on Visual Analogue Scale (VAS) (0=No vestibular symptom, 10=worst vestibular symptom).
Change in number of Moderate/Severe vestibular symptom days as defined by Bárány Society for participants measured daily from the observational phase compared to baseline between group B1 and B2 | 12 weeks after treatment
  After the start of treatment, participants are required to keep a daily dizziness diary. The definition of moderate and severe vestibular symptoms refers to the Barany Society. Symptoms that have an impact on daily activities but can still be endured are defined as moderate, while symptoms that completely prevent daily activities from being carried out are defined as severe.

SECONDARY OUTCOMES:
The percentage of patients satisfied with medication to evaluate the effectiveness of different treatment in the treatment of VM | Within 48 hours post-dose of medication for group A1 and A2, 12-weeks after treatment for group B1 and B2
  Satisfaction with medication will be measured via 7-point SM scale

IPD SHARING:
Plan to Share IPD: No